CLINICAL TRIAL: NCT02991599
Title: Immunogenicity and Persistence of Intramuscular High Dose Recombinant Hepatitis B Vaccine in Methadone Maintenance Treatment Patients in China: a Randomized Controlled Trial
Brief Title: Immunogenicity of Hepatitis B Vaccination in Methadone Maintenance Treatment Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanxi Medical University (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Principal Investigator, Suping Wang, Professor, Shanxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2012ZX10002001003004003
Record Dates: First submitted 2016-12-10; First posted 2016-12-13 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Hepatitis B Vaccine
Keywords: Hepatitis B, Vaccine; Immunogenicity; methadone maintenance treatment; Randomized Controlled Trial
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60 µg dose hepatitis B vaccine (Experimental): 60 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6
  Interventions: Biological: 60 µg dose hepatitis B vaccine
- 20 µg dose hepatitis B vaccine (Experimental): 20 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6
  Interventions: Biological: 20 µg dose hepatitis B vaccine

INTERVENTIONS:
Biological: 60 µg dose hepatitis B vaccine — three-dose, 60 µg per dose
  Arms: 60 µg dose hepatitis B vaccine
Biological: 20 µg dose hepatitis B vaccine — three-dose, 20 µg per dose
  Arms: 20 µg dose hepatitis B vaccine

SUMMARY:
This is a randomized, controlled trial. The study will evaluate the immunogenicity, immune persistence, and safety of 20 µg and 60 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6 in methadone maintenance treatment patients.

DETAILED DESCRIPTION:
Comparison of 2 vaccination strategy against Hepatitis B in patients with Methadone Maintenance Treatment

Intervention:

Arm 1 : 60 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6;

Arm 2 : 20 µg recombinant hepatitis B vaccine with three injections at months 0, 1, and 6.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years at the enrolment
* Serologically negative for hepatitis B surface antigen (HBsAg) and hepatitis B surface antibody (anti-HBs) at enrollment
* Willing to adhere to the study protocol

Exclusion Criteria:

* Being pregnant
* Intolerance or allergy to any component of the vaccine
* Any vaccination during the month preceding enrollment
* Ongoing opportunistic infection
* Liver disease
* Hematological disorder
* Cancer
* Unexplained fever the week before enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suping Wang, Principal Investigator — Shanxi Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shi J, Feng Y, Gao L, Feng D, Yao T, Shi S, Zhang Y, Liang X, Wang S. Immunogenicity and safety of a high-dose hepatitis B vaccine among patients receiving methadone maintenance treatment: A randomized, double-blinded, parallel-controlled trial. Vaccine. 2017 Apr 25;35(18):2443-2448. doi: 10.1016/j.vaccine.2017.03.034. Epub 2017 Mar 23. PMID 28343774

RESULTS

PARTICIPANT FLOW:
Groups:
- IM 20μg Group: Participants received 3 intramuscular injections of 20 μg recombinant hepatitis B vaccine at months 0, 1 and 6.
- IM 60μg Group: Participants received 3 intramuscular injections of 60 μg recombinant hepatitis B vaccine at months 0, 1 and 6.
Period: Overall Study
Arm/Group | IM 20μg Group | IM 60μg Group
Started | 98 | 98
Completed | 60 | 61
Not Completed | 38 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IM 20μg Group | IM 60μg Group | Total
Number analyzed (Participants) | 98 | 98 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (7.5) | 44.0 (7.5) | 43.2 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 41
  Male | 75 | 80 | 155
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han ethnicity | 76 | 83 | 159
  minority ethnicity | 22 | 15 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  China: Urban | 76 | 81 | 157
  China: Rural | 22 | 17 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number and Rate of Participants With Anti-HBs Seroconversion at Month 7
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA（ Chemiluminescent Microparticle Immunoassay ）
  . The accepted protective serum anti-HBs level was ≥10 mIU/ml.
Time Frame: Month 7
Population: 73 and 71 patients in the IM20 and IM60 groups completed the followed-up at months 7.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 73 | 71
Participants | 59 | 62

2. Secondary Outcome: Anti-HBs Concentration at Month 7
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA（ Chemiluminescent Microparticle Immunoassay ）
Time Frame: Month 7
Population: 73 and 71 patients in the IM20 and IM60 groups completed the followed-up at months 7 .
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 73 | 71
mIU/mL | 630.4 [157.7 to 1103.0] | 742.9 [187.0 to 1298.9]

3. Secondary Outcome: Anti-HBs Concentration at Month 12
Description: as for outcome 2
Time Frame: Month 12
Population: 60 and 61 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 60 | 61
mIU/mL | 125.9 [49.9 to 202.0] | 182.2 [97.7 to 266.6]

4. Secondary Outcome: Number and Rate of Participants With Anti-HBs Seroconversion at Month 12
Description: as for outcome 1
Time Frame: Month 12
Population: 60 and 61 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 60 | 61
Participants | 41 | 43

5. Secondary Outcome: Occurrence of Adverse Events After Vaccination
Description: Occurrence of adverse reactions within 7 days after vaccination with the hepatitis B vaccine
Time Frame: Within 7 days after the vaccination, at Month 0, 1, and 6
Population: 196 patients were enrolled and randomized,195 patients received the first dose, 1 patients declined in IM60 group.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 98 | 97
Participants | 7 | 8

6. Secondary Outcome: Occurrence of Adverse Events After Vaccination
Description: Occurrence of adverse reactions within 28 days after vaccination with the hepatitis B vaccine
Time Frame: Within 28 days after the vaccination, at Month 0, 1, and 6
Population: 196 patients were enrolled and randomized,195 patients received the first dose, 1 patients declined in IM60 group.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 98 | 97
Participants | 2 | 3

7. Other Pre Specified Outcome: Number and Rate of Participants With Anti-HBs High-level Response at Month 7
Description: The measurements of anti-HBs antibodies were determined quantitatively by CMIA. and anti-HBs concentrations ≥100 mIU/ml were high-level response.
Time Frame: Month 7
Population: 73 and 71 patients in the IM20 and IM60 groups completed the followed-up at months 7.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 73 | 71
Participants | 31 | 40

8. Other Pre Specified Outcome: Number and Rate of Participants With Anti-HBs High-level Response at Month 12
Description: as for outcome 7
Time Frame: Month 12
Population: 60 and 61 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 60 | 61
Participants | 13 | 20

9. Secondary Outcome: Anti-HBs Concentration at Month 18
Description: as for outcome 2
Time Frame: Month 18
Population: 47 and 43 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 47 | 43
mIU/mL | 382.2 [196.3 to 960.7] | 490.5 [72.4 to 1053.4]

10. Secondary Outcome: Number and Rate of Participants With Anti-HBs Seroconversion at Month 18
Description: as for outcome 1
Time Frame: Month 18
Population: 47 and 43 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 47 | 43
Participants | 29 | 29

11. Other Pre Specified Outcome: Number and Rate of Participants With Anti-HBs High-level Response at Month 18
Description: as for outcome 7
Time Frame: Month 18
Population: 47 and 43 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 47 | 43
Participants | 9 | 14

12. Secondary Outcome: Anti-HBs Concentration at Month 30
Description: as for outcome 2
Time Frame: Month 30
Population: 46 and 42 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 46 | 42
mIU/mL | 239.9 [119.3 to 599.1] | 306.4 [60.2 to 579.3]

13. Secondary Outcome: Number and Rate of Participants With Anti-HBs Seroconversion at Month 30
Description: as for outcome 1
Time Frame: Month 30
Population: 46 and 42 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 46 | 42
Participants | 20 | 25

14. Secondary Outcome: Anti-HBs Concentration at Month 42
Description: as for outcome 2
Time Frame: Month 42
Population: 45 and 40 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 45 | 40
mIU/mL | 88.6 [12.4 to 170] | 97.7 [17.5 to 186.6]

15. Secondary Outcome: Number and Rate of Participants With Anti-HBs Seroconversion at Month 42
Description: as for outcome 1
Time Frame: Month 42
Population: 45 and 40 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 45 | 40
Participants | 14 | 20

16. Other Pre Specified Outcome: Number and Rate of Participants With Anti-HBs High-level Response at Month 30
Description: as for outcome 7
Time Frame: Month 30
Population: 46 and 42 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 46 | 42
Participants | 6 | 11

17. Other Pre Specified Outcome: Number and Rate of Participants With Anti-HBs High-level Response at Month 42
Description: as for outcome 7
Time Frame: Month 42
Population: 45 and 40 patients in the IM20 and IM60 groups completed the followed-up at months 12.
Measure: Count of Participants; unit: Participants
Arm/Group | IM 20μg Group | IM 60μg Group
Number analyzed (Participants) | 45 | 40
Participants | 4 | 8

ADVERSE EVENTS:
Arm/Group | IM 20μg Group | IM 60μg Group
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/97
Other Adverse Events (participants affected / at risk) | 7/98 | 8/97
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IM 20μg Group (N=98) | IM 60μg Group (N=97)
pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Erythema (Skin and subcutaneous tissue disorders) | 5 | 5
Edema (Skin and subcutaneous tissue disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No